CLINICAL TRIAL: NCT05601141
Title: Pituitary Diseases in Modena Population: Clinical and Epidemiological Data Register of Pituitary Patients Attending the Unit of Endocrinology of Azienda Ospedaliero-Universitaria of Modena (DataPit)
Brief Title: Clinics and Epidemiology of Pituitary Diseases in Modena Area Population
Acronym: DataPit
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Principal Investigator, Vincenzo Rochira, MD, PhD - Associate Professor of Endocrinology, Azienda Ospedaliero-Universitaria di Modena
Other Study IDs: 289/2021
Record Dates: First submitted 2022-10-24; First posted 2022-11-01 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Pituitary
MeSH Terms: conditions — Pituitary Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is an observational, longitudinal, single-center study.

The study is divided in two phases:

* FIRST PHASE (retrospective): registration of all patients affected by pituitary disorders followed at the Unit of Endocrinology of Azienda Ospedaliero-Universitaria of Modena
* SECOND PHASE (prospective): enrollment of all patients affected by pituitary disorders who attend the Unit of Endocrinology of the Azienda Ospedaliero-Universitaria of Modena.

An anonymized database will be created to collect the data of the patients. In particular, the data collected for each patient will include: personal data, data relating to pituitary pathology, symptoms at diagnosis, physical examination, radiological imaging, visual field data, data on surgical intervention, data on histological examination, biohumoral examinations, hormone tests, densitometric data, data on replacement therapies, medical therapies or other pharmacological therapies, data on comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* subjects affected by pituitary disorders who attended Unit of Endocrinology of Azienza Ospedaliero-Universitaria di Modena

Exclusion Criteria:

* subjects under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by pituitary disorders who attended Unit of Endocrinology of Azienza Ospedaliero-Universitaria di Modena
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2031-10-24 (Estimated); Study Completion 2031-10-24 (Estimated)

PRIMARY OUTCOMES:
Characterization of pituitary patients | 10 years
  The primary aim of the study is to characterize subjects with pituitary disease by collecting anamnestic, clinical, biohumoral, radiological data, and data related to the treatment approach, in terms of surgery, medical therapies and/or hormone replacement therapies.

SECONDARY OUTCOMES:
Management of pituitary patients | 10 years
  The second aim is to integrate these data with current knowledge, in order to improve the clinical-diagnostic-therapeutic management of patients suffering from pituitary diseases, as well as to identify risk factors for the development of the disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Unit of Endocrinology of Azienza Ospedaliero-Universitaria di Modena, Modena, Modena, Italy

REFERENCES:
- [Background] Freda PU, Beckers AM, Katznelson L, Molitch ME, Montori VM, Post KD, Vance ML; Endocrine Society. Pituitary incidentaloma: an endocrine society clinical practice guideline. J Clin Endocrinol Metab. 2011 Apr;96(4):894-904. doi: 10.1210/jc.2010-1048. PMID 21474686
- [Background] Molitch ME. Management of incidentally found nonfunctional pituitary tumors. Neurosurg Clin N Am. 2012 Oct;23(4):543-53. doi: 10.1016/j.nec.2012.06.003. Epub 2012 Jul 31. PMID 23040742
- [Background] Vasilev V, Rostomyan L, Daly AF, Potorac I, Zacharieva S, Bonneville JF, Beckers A. MANAGEMENT OF ENDOCRINE DISEASE: Pituitary 'incidentaloma': neuroradiological assessment and differential diagnosis. Eur J Endocrinol. 2016 Oct;175(4):R171-84. doi: 10.1530/EJE-15-1272. Epub 2016 Apr 11. PMID 27068689
- [Background] Buurman H, Saeger W. Subclinical adenomas in postmortem pituitaries: classification and correlations to clinical data. Eur J Endocrinol. 2006 May;154(5):753-8. doi: 10.1530/eje.1.02107. PMID 16645024
- [Background] Tresoldi AS, Carosi G, Betella N, Del Sindaco G, Indirli R, Ferrante E, Sala E, Giavoli C, Morenghi E, Locatelli M, Milani D, Mazziotti G, Spada A, Arosio M, Mantovani G, Lania AGA. Clinically Nonfunctioning Pituitary Incidentalomas: Characteristics and Natural History. Neuroendocrinology. 2020;110(7-8):595-603. doi: 10.1159/000503256. Epub 2019 Sep 13. PMID 31525736
- [Background] Mai K, Fassnacht M, Fuhrer-Sakel D, Honegger JB, Weber MM, Kroiss M. The Diagnosis and Management of Endocrine Side Effects of Immune Checkpoint Inhibitors. Dtsch Arztebl Int. 2021 Jun 11;118(Forthcoming):389-96. doi: 10.3238/arztebl.m2021.0143. Online ahead of print. PMID 33724917